CLINICAL TRIAL: NCT07154693
Title: Wound Healing Following Tooth Extraction and Ridge Preservation Using Resorbable Non-ceramic Calcium Apatite Granules in Type I Bovine Collagen Plugs (OsteoGen®)
Brief Title: Wound Healing Following Tooth Extraction and Ridge Preservation Using OsteoGen®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00001531
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Tooth Extraction
Keywords: Wound healing; Vital bone; Mineralized freeze-dried bone allograft (FDBA); Demineralized freeze-dried bone allograft (DFDBA); Ridge preservation

STUDY DESIGN:
Intervention Model Description: Single-study-site parallel-arm randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blind to the material used for their bone graft. Histomorphometric examiners will be blinded when the bone cores are evaluated for % vital bone, % residual graft and % CT/other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Osteogen Test Group (Active Comparator): A synthetic calcium apatite material combined with Type 1 bovine collagen (in a sponge-like product) called "OsteoGen plug®
  Interventions: Device: OsteoGen Plug
- FDBA/DFDBA Control Group (Active Comparator): A synthetic calcium apatite material combined with Type 1 bovine collagen (in a sponge-like product) called "OsteoGen plug®
  Interventions: Device: Combination 70% FDBA and 30% DFDBA

INTERVENTIONS:
Device: Combination 70% FDBA and 30% DFDBA — A combination freeze-dried bone allograft consisting of 70% mineralized FDBA and 30% demineralized FDBA
  Other Names: FDBA/DFDBA
  Arms: FDBA/DFDBA Control Group
Device: OsteoGen Plug — A synthetic calcium apatite material combined with Type 1 bovine collagen (in a sponge-like product)
  Other Names: Osteogen
  Arms: Osteogen Test Group

SUMMARY:
After the removal of a tooth, a bone graft is often placed in the socket to try to keep the volume of bone that was there when the tooth was present so that the bone does not "shrink". The bone graft is sometimes kept in place with a small piece of material over the top of the tooth socket and with stitches. This procedure is called "Ridge Preservation". Many different materials are used for ridge preservation including bone allografts (bone grafts derived from a human tissue donor), bone xenografts (bone grafts derived from species other than humans, such as cows and pigs), and synthetic materials that are similar in structure to bone (such as calcium apatite). The bone allograft and the calcium apatite product used in this study are Food and Drug Administration (FDA) approved.

This study will compare the two methods used to see how much new bone formation there is inside the tooth socket at about 16 weeks of healing after ridge preservation with a calcium apatite/collagen sponge versus an allograft.

DETAILED DESCRIPTION:
At the end of this study the researchers hope to learn the following: How much new bone formation occurs inside the tooth socket at approximately 16 weeks of healing after ridge preservation with calcium apatite/collagen versus allograft.

This will be done by examining the bone retrieved from the implant site during the placement of the implant at study visit #5. This bone is normally removed during the drilling of the implant site and discarded as part of standard care. As part of this study, the bone specimen will be removed as normal but will not be discarded; instead, it will be analyzed for the purpose of this research study.

At the end of this study the researchers hope to learn the following: How much new bone formation occurs inside the tooth socket at approximately 16 weeks of healing after ridge preservation with calcium apatite/collagen versus allograft.

The study team will do this by examining the bone retrieved from the implant site during the placement of the implant at study visit #5. This bone is normally removed during the drilling of the implant site and discarded as part of standard care. As part of this study, the bone specimen will be removed as normal but will not be discarded; instead, it will be analyzed for the purpose of this research study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 to 89
* One tooth, excluding molars, that has been identified by dental faculty as requiring a single tooth extraction
* A dental implant is indicated and treatment planned to replace the missing tooth
* Site has adequate restorative space for a dental implant-retained restoration
* Site has at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Site has a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and nonpregnant women of child-bearing potential.
* Patients are nonsmokers or former smokers. Current smokers may be included if they smoke <10 cigarettes per day (less than or equal to 10 cigarettes per day)

Exclusion Criteria:

* Patient allergic to bovine-derived collagen products, Bacitracin, Gentamicin, Polymyxin
* Patients who will not cooperate with the follow-up schedule.
* Patients will not be entered who are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period (as confirmed verbally; an over-the-counter pregnancy test will be provided if pregnancy status is unknown or suspected).

  * Patients who become pregnant during the study will be withdrawn and standard care will be delivered.
* Smokers who smoke >10 cigarettes per day (more than 10 cigarettes per day)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Vital Bone formation | 16 weeks
  Bone cores will be evaluated histomorphometrically for the primary outcome: % vital bone formation

SECONDARY OUTCOMES:
Percentage of Residual Graft Material | 16 weeks
  Determine percentage of residual graft remaining at time of implant placement
Percentage of CT/other | 16 weeks
  Determine the percentage of residual graft and connective tissue or other tissue at the time of implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mealey, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio School of Dentistry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be thoroughly de-identified and will not be traceable to a specific study participant. If the results of this study are reported in medical journals or at meetings, you will not be identified.
Supporting Information: Study Protocol, SAP
Time Frame: The investigators plan to publish the data once the study is complete and data analysis has occurred. Summary results will also be reported on ClinicalTrials.gov at least one year after primary completion date is reached.